CLINICAL TRIAL: NCT03021395
Title: Efficacy of Decitabine in Clearance of MRD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016007（Decitabine）
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2019-03

CONDITIONS: AML
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD-positive (Experimental): MRD-positive patients receive Decitabine regimen.
  Interventions: Drug: Decitabine
- MRD-negative (No Intervention): MRD-negative patients receive no intervention.

INTERVENTIONS:
Drug: Decitabine — Decitabine at a dose of 20mg/㎡/d on day 1-5.
  Arms: MRD-positive

SUMMARY:
In this open-label, prospective clinical trial, the investigators enrolled acute myeloid leukemia (AML) patients after consolidation therapy. Patients with minimal residual disease (MRD) receive decitabine treatment if patients do not receive stem cell transplantation. The MRD clearance rate is the primary outcome to measure the efficacy of decitabine regimen.

DETAILED DESCRIPTION:
In this open-label, prospective clinical trial, acute myeloid leukemia (AML) patients after consolidation therapy are enrolled. Patients with minimal residual disease (MRD) after consolidation therapy receive decitabine treatment if patients do not receive stem cell transplantation. The treatment regimen includes three course of decitabine regimen at a dose of 20mg/m² on day1-5. The MRD clearance rate is the primary outcome to measure the efficacy of decitabine regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 14 to 55 years old;
2. Patients that meet the diagnostic criteria(WHO 2008 criteria) of AML after consolidation regimen.
3. Patients who had received induction and consolation therapy and reached CR.
4. ECOG score of ≤ 2;
5. Patients with eligible laboratory examination including liver,renal and heart function.
6. Adult patients are willing to participate in the study and sign the informed consent by themselves or by their immediate family. Patients under 18 years old willing to participate should have their legal guardians sign the informed consent.

Exclusion Criteria:

1. Secondary leukemia.
2. Patients had other tumor at active stage or had received radiotherapy or chemotherapy in the last 6 months due to other tumor.
3. Patients with other blood diseases(for example, haemophiliacs) are excluded.However, undiagnosed MDS or MPD patients are included.
4. Acute panmyelosis with myelofibrosis and myeloid sarcoma patients;
5. With BCR-ABL fusion gene;
6. Pregnant or lactating women;
7. With ineligible renal or liver function;
8. With active cardiovascular disease;
9. Severe infection disease including uncured tuberculosis pulmonary aspergillosis;
10. AIDS;
11. Patients had central nervous system involvement when they were diagnosed as AML.
12. Patients with epilepsy or dementia or other mental disease who couldn't understand or follow the research.
13. Drugs, medical, mental or social situation may distract patients from following the research or being evaluated the results.
14. Patients with other factors which were considered unsuitable to participate in the study by the investigators.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
MRD Clearance Rate | Within 6 months after decitabine treatment
  MRD Clearance Rate is defined as the ratio patients that transform from MRD-positive to MRD-negative after treatment in all of the MRD-positive patients.

SECONDARY OUTCOMES:
Non-relapse Mortality | Within 5 years after treatment
Overall Survival Rate (OS) | Within 5 years after treatment
Cumulative incidence of relapse | Within 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No